CLINICAL TRIAL: NCT03770923
Title: Clinical Study Evaluating the Effect of Histamine 1 Receptor Antagonist and Leukotreine Receptor Antagonist on Patients With Rheumatoid Arithritis
Brief Title: Effect of Some Drugs on Rheumatoid Arithritis Activity
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rheumatoid Arithritis
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — rupatadine; montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No intervention (No Intervention): No intervention
- Rupatadine (Active Comparator): Rupatadine 10 mg once daily.
  Interventions: Drug: Rupatadine
- Montelukast (Active Comparator): Montelukast 10 mg daily
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Rupatadine — Rupatadine 10 mg daily
  Arms: Rupatadine
Drug: Montelukast — Montelukast 10 mg daily
  Arms: Montelukast

SUMMARY:
Effect of Some Drugs on Rheumatoid Arithritis Activity.

DETAILED DESCRIPTION:
The study aims at evaluating the effect of Some Drugs on Rheumatoid Arithritis Activity.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis

Exclusion Criteria:

* liver or renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
se level of IL-17 | 6 months
  change in level of IL-17

CONTACTS AND LOCATIONS:
Overall Officials: Sahar k Hegazy, Prof, Principal Investigator — Head of Clinical Pharmacy Department; Tarek M Mostafa, Prof, Study Director — Clinical pharmacy Department- Tanta University; Salwa E Abd El-Ghany, Prof, Study Chair — Rheumatology Dept. - Tanta University; Fedaa AK Kotkata, Msc, Study Chair — Clinical pharmacy Department-Tanta University
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mostafa TM, Hegazy SK, El-Ghany SEA, Kotkata FAE. Comparative study evaluating antihistamine versus leukotriene receptor antagonist as adjuvant therapy for rheumatoid arthritis. Eur J Clin Pharmacol. 2021 Dec;77(12):1825-1834. doi: 10.1007/s00228-021-03181-2. Epub 2021 Jul 4. PMID 34218304